CLINICAL TRIAL: NCT04264104
Title: Effect of Nervous System Mobilization on Athletes' Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-CED/2019
Record Dates: First submitted 2020-02-06; First posted 2020-02-11 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2020-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose neural mobilization (Experimental): Four series of 10 repetitions of neural mobilization targeting the tibial nerve.
  Interventions: Other: neural mobilization
- High dose neural mobilization (Active Comparator): Eight series of 10 repetitions of neural mobilization targeting the tibial nerve.
  Interventions: Other: neural mobilization

INTERVENTIONS:
Other: neural mobilization — This is a type of mobilization that uses a specific combination of joint movements

SUMMARY:
This study aims to compare the effects of two diferente doses of nervous system mobilization on athletes performance.

DETAILED DESCRIPTION:
It is anticipated that 60 athletes will be randomly allocated to receive either 4x10 (n=30) or 8x10 (n=30) repetitions of neural mobilization .

Data on flexibility (knee extension test) and lower limb strength and motor control (hop tests and vertical jump test) will be collected at baseline and after the neural mobilization.

Statistical analysis will be performed using a mixed-methods ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy athletes

Exclusion Criteria:

* Nerve damage
* Arthritis
* Tumors
* Vascular conditions
* Spinal cord injuries
* Any sistemic condition
* Surgery in the past 6 months
* Injury in the last 3 months
* A knee angle of <10º

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Single Leg Hop Test | Baseline
  Participants are asked to perform one single unipedal jump and the jump width is measured.
Single Leg Hop Test | Up to 1 hour after baseline
  Participants are asked to perform one single unipedal jump and the jump width is measured.
Crossover Test | Baseline
  Participants are asked to jump as far as possible on a single leg three consecutive times, without losing balance and landing firmly. The total width of the 3 consecutive jumps is measured.
Crossover Test | Up to 1 hour after baseline
  Participants are asked to jump as far as possible on a single leg three consecutive times, without losing balance and landing firmly. The total width of the 3 consecutive jumps is measured.

SECONDARY OUTCOMES:
6-meter Time Hop Test | Baseline
  The aim is to jump as fast as possible on a single leg over a distance of 6 meters, without losing balance and landing firmly. The time taken to perform this test is the measure of interest.
6-meter Time Hop Test | Up to 1 hour after baseline
  The aim is to jump as fast as possible on a single leg over a distance of 6 meters, without losing balance and landing firmly. The time taken to perform this test is the measure of interest.
Vertical Jump test | Baseline
  Participants are asked to jump upwards and the height jumped is measured.
Vertical Jump test | Up to 1 hour after baseline
  Participants are asked to jump upwards and the height jumped is measured.
Knee extension test | Baseline
  Participants are in a prone position, hip at 90º flexion and knee extension is performed. The measure of interest is the knee extension angle.
Knee extension test | Up to 1 hour after baseline
  Participants are in a prone position, hip at 90º flexion and knee extension is performed. The measure of interest is the knee extension angle.

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Silva, Principal Investigator — Aveiro University
Locations (1):
- basketball teams at Aveiro region, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No